CLINICAL TRIAL: NCT01205893
Title: Study to Confirm the Safety and Efficacy of the Reducer on Patients With Refractory Angina
Brief Title: Coronary Sinus Reducer for Treatment of Refractory Angina - COSIRA
Acronym: COSIRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shockwave Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #REDCLN-178
Record Dates: First submitted 2010-09-13; First posted 2010-09-21 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Refractory Angina
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reducer (Experimental): Implant Reducer
  Interventions: Device: Neovasc Reducer
- Control (Sham Comparator): No treatment
  Interventions: Device: Control

INTERVENTIONS:
Device: Neovasc Reducer — Implantation of the Reducer
  Arms: Reducer
Device: Control — Control - No device implanted
  Arms: Control

SUMMARY:
The purpose of this study is to determine if the Reducer is safe and effective in treating the symptoms of refractory angina in patients that suffer from refractory angina who demonstrate reversible ischemia.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is older than 18 years of age
2. Symptomatic CAD with chronic refractory angina pectoris classified as Canadian Cardiovascular Society grade III or IV despite attempted optimal medical therapy for thirty days prior to screening
3. Patient has limited treatment options for revascularization by coronary artery bypass grafting or by percutaneous coronary intervention
4. Evidence of reversible ischemia that is attributable to the left coronary arterial system by Dobutamine Echo
5. Left ventricular ejection fraction greater than 25%
6. Male or non-pregnant female (NB: Females of child bearing potential must have a negative pregnancy test)
7. Patient understands the nature of the procedure and provides written informed consent prior to enrollment
8. Patient is willing to comply with specified follow-up evaluation and can be contacted by telephone

Exclusion Criteria:

1. Recent (within three months) acute coronary syndrome
2. Recent (within six months) successful PCI or CABG
3. Unstable angina (recent onset angina, crescendo angina, or rest angina with ECG changes) during the thirty days prior to screening
4. De-compensated congestive heart failure (CHF) or hospitalization due to CHF during the three months prior to screening
5. Life threatening rhythm disorders or any rhythm disorders that would require placement of an internal defibrillator and or pacemaker
6. Severe chronic obstructive pulmonary disease (COPD) as indicated by a forced expiratory volume in one second that is less than 55% of the predicted value
7. Patient cannot undergo exercise tolerance test (bicycle) for reasons other than refractory angina
8. Severe valvular heart disease
9. Patient with pacemaker or defibrillator electrode in the right atrium, right ventricle, or coronary sinus
10. Patient having undergone tricuspid valve replacement or repair
11. Chronic renal failure (serum creatinine >2 mg/dL), including patients on chronic hemodialysis
12. Moribund patients, or patients with comorbidities limiting life expectancy to less than one year
13. Contraindication to required study medications that cannot be adequately controlled with pre-medication
14. Known allergy to stainless steel or nickel
15. Contraindication to having an MRI performed (NB: Cardiac MRI subset patients only)
16. Currently enrolled in another investigational device or drug trial that has not completed the primary endpoint or that clinically interferes with the current study endpoints
17. Mean right atrial pressure higher than or equal to 15 mmHg
18. Patient with anomalous or abnormal CS as demonstrated by angiogram. Abnormality defined as:

Abnormal CS anatomy (e.g., tortuosity, aberrant branch, persistent left SVC) and/or; CS diameter at the site of planned reducer implantation less than 9.5 mm or greater than 13 mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2010-09; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Canadian Cardiovascular Society Angina Score | 6 months
  A decrease of two or more Canadian Cardiovascular Society Angina Score grades from baseline to six-month post-procedural evaluation in Reducer and Control groups

SECONDARY OUTCOMES:
Technical success | 24 hours
  Successful delivery and deployment of the Reducer to the intended site as assessed by the investigator
Procedural success | 24 hours
  Technical success and the absence of acute need for clinically-driven intervention to address an Adverse or Serious Adverse Device Effect prior to hospital discharge
Periprocedural Serious Adverse Event: | 30 days
  A composite of death, myocardial infarction, cardiac tamponade, clinically-driven re-dilation of a failed Reducer, life-threatening arrhythmia, and respiratory failure through 30 days post-procedure in the Reducer group.
Periprocedural Serious Adverse Event | 30 days
  A composite of death, myocardial infarction, cardiac tamponade, life-threatening arrhythmia, and respiratory failure through 30 days post-procedure in the control group.
Major Adverse Events | 6 months
  A composite of cardiac death, major stroke, and myocardial infarction in the Reducer and Control groups through hospital discharge, and at six-month post-procedural evaluations.
Canadian Cardiovascular Society Angina Score | 6 months
  A decrease one or more Canadian Cardiovascular Society Angina Score grades from baseline to six-month post-procedural evaluation in Reducer and Control groups
Dobutamine Echo Wall Motion Score Index | 6 months
  Wall motion score index in both the Reducer and control groups at baseline and six-month post-procedural evaluation
Seattle Angina Questionnaire Score | 6 months
  Seattle Angina Questionnaire in the Reducer and Control groups at baseline and six-month post-procedural evaluation
Exercise Tolerance Testing | 6 months
  Exercise Tolerance Testing in the Reducer and Control groups at baseline and six-month post-procedural evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Verheye, MD, Principal Investigator — ZNA Middelheim Hospital
Locations (11):
- Belgium (2):
  - ZNA Middelheim Hospital, Antwerp
  - Ziekenhuis Oost-Limburg, Genk
- Canada (2):
  - Ottawa Heart Institute, Ottawa, Ontario
  - Montreal Heart Institute, Montreal, Quebec
- Rigshospitalet, Copenhagen, Denmark
- UMC Utrecht, Utrecht, Netherlands
- Central Hospital Kristianstad, Kristianstad, Sweden
- United Kingdom (4):
  - Royal Infirmary of Bradford, Bradford
  - Royal Infirmary of Edinburgh, Edinburgh
  - King College Hospital, London
  - Royal Brompton Hospital, London

REFERENCES:
- [Derived] Jolicoeur EM, Verheye S, Henry TD, Joseph L, Doucet S, White CJ, Edelman E, Banai S. A novel method to interpret early phase trials shows how the narrowing of the coronary sinus concordantly improves symptoms, functional status and quality of life in refractory angina. Heart. 2021 Jan;107(1):41-46. doi: 10.1136/heartjnl-2020-316644. Epub 2020 Jul 21. PMID 32719097
- [Derived] Verheye S, Jolicoeur EM, Behan MW, Pettersson T, Sainsbury P, Hill J, Vrolix M, Agostoni P, Engstrom T, Labinaz M, de Silva R, Schwartz M, Meyten N, Uren NG, Doucet S, Tanguay JF, Lindsay S, Henry TD, White CJ, Edelman ER, Banai S. Efficacy of a device to narrow the coronary sinus in refractory angina. N Engl J Med. 2015 Feb 5;372(6):519-27. doi: 10.1056/NEJMoa1402556. PMID 25651246
- [Derived] Jolicoeur EM, Banai S, Henry TD, Schwartz M, Doucet S, White CJ, Edelman E, Verheye S. A phase II, sham-controlled, double-blinded study testing the safety and efficacy of the coronary sinus reducer in patients with refractory angina: study protocol for a randomized controlled trial. Trials. 2013 Feb 15;14:46. doi: 10.1186/1745-6215-14-46. PMID 23413981